CLINICAL TRIAL: NCT01138722
Title: Pathologic Effects of Neoadjuvant Radiation Therapy in Operable Early Stage Lung Cancer
Brief Title: Predicting Cell Death by Radiation Therapy in Early Stage Non-small Cell Lung Cancer: a Prospective Translational Trial
Acronym: PEARL-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment rate.
Sponsor: University Hospital, Ghent (Other)
Collaborators: Nationaal Kankerplan (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010/204; LONG 10-01 (Other: University Hospital Ghent)
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Early Stage Non-small Cell Lung Cancer
Keywords: early stage non-small cell lung cancer; hypofractionated radiation therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: hypofractionated radiation therapy followed by surgery — hypofractionated radiation therapy followed by surgery

SUMMARY:
Surgical resection with mediastinal lymph node sampling is currently the therapy of choice for early stage (I-II) non-small cell lung cancer (NSCLC). Selected patients unwilling or unable to tolerate surgery are referred for so-called 'curative' high dose radiotherapy. This has shown to result in a long term local disease control rate and a high cancer specific survival.

The current trial addresses the relationship between blood and tissue biomarkers, bio-imaging and pathology in patients with early stage NSCLC treated with hypofractionated radiation therapy and surgery.

ELIGIBILITY:
Inclusion Criteria:

* Proof of cT1a/b - 2a/b N0M0 NSCLC
* Informed Consent signed
* Resectable tumour
* Operable patient
* > 18 years old
* men and women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
pathological effects of hypofractionated radiation therapy | at 2 years
  To describe the pathological effects of hypofractionated radioation therapy (RT) and to address the relationship with blood and tissue biomarkers and bio-imaging.

SECONDARY OUTCOMES:
clinical response rate | from 2 to 5 years
the accuracy of clinical mediastinal staging | from 2 to 5 years
the complication rate | from 2 to 5 years
local, regional or distant failure | from 2 to 5 years
progression free survival | from 2 to 5 years
disease specific overall survival | from 2 to 5 years
overall survival | from 2 to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan Van Meerbeeck, MD, PhD, Principal Investigator — University Hospital Ghent, Belgium
Locations (2):
- Belgium (2):
  - University Hospital Antwerp, Antwerp
  - University Hospital Ghent, Ghent

REFERENCES:
- See also: website of University Hospital Ghent — http://www.uzgent.be